CLINICAL TRIAL: NCT02435888
Title: Accuracy and Agreement of Predictive Equations for Resting Energy Expenditure Among Overweight Patients With Polycystic Ovary Syndrome
Brief Title: Predictive Equations for Resting Energy Expenditure
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Professor, Department of Surgery, School of Medicine, Federal University of Minas Gerais
Other Study IDs: ETIC 0244.0.0203.000-10
Record Dates: First submitted 2015-05-03; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Resting energy expenditure; Predictive equations; Overweight
MeSH Terms: conditions — Polycystic Ovary Syndrome; Overweight

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Polycystic ovary syndrome

SUMMARY:
Predictive equations are the main clinical tool for determining resting energy expenditure (REE). Thus, it is important to investigate the accuracy and agreement of these equations in different populations and context of diseases. The purpose of this study is to investigate the accuracy and agreement of predictive equations of REE in overweight women with polycystic ovary syndrome (PCOS). The REE of all participants was measured (mREE) by means of indirect calorimetry and predicted (pREE) through ten equations basing on the anthropometric parameters (Harris & Benedict, WHO/FAO/UNU including weight, WHO/FAO/UNU including weight and height, Owen, Mifflin-St. Jeor, Institute of Medicine, Ireton-Jones, Müeller, De Luis and Lazzer).

ELIGIBILITY:
Inclusion Criteria:

* Women treated in an endocrinology centre specialising in hyperandrogenism at the university hospital of University Federal of Minas Gerais (Belo Horizonte, Minas Gerais, Brazil)
* The patients were of reproductive age (range: 18-45 years)
* were overweight or obese (Body mass index ≥ 25.0 kg/m2) and
* signed an informed consent statement

Exclusion Criteria:

* Women who were pregnant,
* were lactating,
* had a diagnosis of hypothyroidism or hyperthyroidism or
* had high physical activity levels were excluded from the sample.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Polycystic ovary syndrome patients, as defined according to the Rotterdam criteria (ESHRE/ASMR, 2004): the presence of at least two of the following factors: chronic anovulation, clinical or biochemical signs of hyperandrogenism and presence of polycystic ovaries;
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Accuracy and agreement of predictive equations of resting energy expenditure | Six month

SECONDARY OUTCOMES:
Comparison and correlation between the resting energy expenditure measured by means of indirect calorimetry and predicted through equations. | Six month

CONTACTS AND LOCATIONS:
Overall Officials: Adaliene VM Ferreira, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- UFMG Hospital, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Derived] Rodrigues AMDS, Costa ABP, Campos DL, Silva MPS, Candido AL, Santos LCD, Ferreira AVM. Low validity of predictive equations for calculating resting energy expenditure in overweight and obese women with polycystic ovary syndrome. J Hum Nutr Diet. 2018 Apr;31(2):266-275. doi: 10.1111/jhn.12498. Epub 2017 Aug 8. PMID 28791776